CLINICAL TRIAL: NCT00730925
Title: A Phase II Single-arm Trial of BIBW 2992 in Demographically and Genotypically Selected NSCLC
Brief Title: Single-arm Trial of BIBW 2992 (Afatinib) in Demographically and Genotypically Selected NSCLC Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.41; 2008-001546-67 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-06-30; First posted 2008-08-08 (Estimated); Results first posted 2013-10-23 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib; Paclitaxel

ARMS (2):
- BIBW 2992 (Experimental): patient to receive tablets of BIBW 2992 once a day, starting at high dose until progression of the disease
  Interventions: Drug: BIBW2992
- BIBW 2992 + paclitaxel (Experimental): patient whose disease progressed on treatment with BIBW 2992 monotherapy to receive tablet of BIBW 2992 once a day in combination with i.v. paclitaxel 3 weekly
  Interventions: Drug: BIBW2992 + paclitaxel

INTERVENTIONS:
Drug: BIBW2992 — tablet BIBW high dose
  Arms: BIBW 2992
Drug: BIBW2992 + paclitaxel — tablet BIBW 2992 in combination with i.v. paclitaxel 3 weekly
  Arms: BIBW 2992 + paclitaxel

SUMMARY:
The primary objective of this open-label, single arm Phase II trial is to explore the efficacy of BIBW 2992 defined by the objective response rate (CR, PR) as determined by the RECIST criteria, in patients with advanced NSCLC Stage IIIB or IV whose tumours harbour activating mutations within exon 18 to exon 21 of the EGFR receptor, in patients with mutations in the HER2/neu receptor and in patients with EGFR FISH positive tumours with no EGFR mutations.

ELIGIBILITY:
Inclusion criteria:

1. patients with pathologically confirmed diagnosis of NSCLC stage IIIB/IV adeno- or bronchoalveolar carcinoma (BAC)
2. non smokers patients or patients having smoked less than 15 pack years and who stopped smoking for at least one year before diagnosis (except for patients with her2-neu mutation)
3. presence of activating mutation(s) in exon 18 to exon 21 of the EGFR or HER2-neu-receptor confirmed by direct DNA sequencing of NSCLC tumor tissue or increased copy number of the EGFR gene as determined by FISH analysis
4. prior treatment up to 3 lines of chemotherapy except for HER2-neu patients (no restrictions) no prior EGFR TKI therapy for EGFR mutation negative and FISCH positive patients
5. patients with at least one tumor lesion that can accurately be measured by CTscan or MRI in at least one dimension with long diameter to be recorded as > or equal to 20 mm using conventional techniques or > or equal to 10 mm with spiral CT scan
6. male or female patient aged above or equal to 18 years
7. life expectancy of at least 3 months
8. written informed consents that is consistent with ICH-GCP guidelines
9. ECOG performance score 0, 1 or 2

Exclusion criteria:

1. more than 3 prior cytotoxic chemotherapy treatment regimen for relapsed or metastatic NSCLC, except for patients with HER2-neu mutations who may have received any prior therapy
2. Any chemo-, hormone- or immunotherapy within the past 4 weeks or within less than 4 half-lives of the previous drug prior to treatment with the trial drug and/or persistence of toxicities of prior anticancer therapies which are deemed to be clinically relevant
3. brain metastases which are symptomatic; patients with treated asymptomatic brain metastases are eligible with stable brain disease for at least 4 weeks without requirement for steroids or anti-epileptic therapy
4. significant or recent acute gastrointestinal disorders with diarrhea as a major symptom e.g. Crohn's disease, malabsorption or CTCAE Grade > 2 diarrhea of any etiology at baseline
5. patients who have any other life-threatening illness or organ system dysfunction, which in the opinion of the investigator, would either compromise patient safety or interfere with the evaluation of the safety of the test drug
6. other malignancies diagnosed within the past 5 years (other than non melanomatous skin cancer and in situ cervical cancer)
7. radiotherapy within the past 2 weeks prior to treatment with the trial drug
8. patients with any serious active infection (i.e., requiring an IV antibiotic, antifungal, or antiviral agents)
9. patients with known HIV, active hepatitis B or active hepatitis C
10. known or suspected active drug or alcohol abuse
11. women of childbearing potential or men who are able to father a child unwilling to use a medically acceptable method of contraception during the trial
12. pregnancy or breast feeding
13. patient unable to comply with the protocol
14. history of clinically significant or uncontrolled cardiac disease, including congestive heart failure, angina, myocardial infarction, arrhythmia, including New York Heart Association (NYHA) functional classification of 3
15. Cardiac left ventricular function with resting ejection fraction of less than 50% measured by multigated blood pool imaging of the heart (MUGA scan) or Echocardiogram.
16. Absolute neutrophil count (ANC) less than 1500/mm³.
17. Platelet count less than 100 000 / mm³.
18. Bilirubin greater than 1.5 mg / dl (>26 µmol / L, SI unit equivalent).
19. Aspartate amino transferase (AST) or alanine amino transferase (ALT) greater than three times the upper limit of normal (if related to liver metastases greater than five times the upper limit of normal).
20. Serum creatinine greater than 1.5 times of the upper normal limit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-06; Primary Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (7):
- Belgium (6):
  - 1200.41.32003 Boehringer Ingelheim Investigational Site, Antwerp
  - 1200.41.32007 Boehringer Ingelheim Investigational Site, Charleroi
  - 1200.41.32001 Boehringer Ingelheim Investigational Site, Jette
  - 1200.41.32011 Boehringer Ingelheim Investigational Site, Leuven
  - 1200.41.32008 Boehringer Ingelheim Investigational Site, Liège
  - 1200.41.32006 Boehringer Ingelheim Investigational Site, Namur
- 1200.41.34001 Boehringer Ingelheim Investigational Site, Badalona (Barcelona), Spain

REFERENCES:
- [Derived] De Greve J, Teugels E, Geers C, Decoster L, Galdermans D, De Mey J, Everaert H, Umelo I, In't Veld P, Schallier D. Clinical activity of afatinib (BIBW 2992) in patients with lung adenocarcinoma with mutations in the kinase domain of HER2/neu. Lung Cancer. 2012 Apr;76(1):123-7. doi: 10.1016/j.lungcan.2012.01.008. Epub 2012 Feb 10. PMID 22325357

RESULTS

PARTICIPANT FLOW:
Groups:
- Afatinib 50mg: Afatinib 50mg film coated tablets were administered once daily as long as they were tolerated by patients, until disease progression (according to the response evaluation criteria in solid tumors)
Period: Overall Study
Arm/Group | Afatinib 50mg
Started | 41
Completed | 0 (On treatment at analysis cut-off date)
Not Completed | 41
Not completed — Progressive Disease | 21
Not completed — Dose reducing Event | 2
Not completed — Other Averse Event | 7
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1
Not completed — Switch to combination therapy | 8
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Best Objective Response
Description: Percentage of participants with best objective response: confirmed complete response (CR) or confirmed partial response (PR) according to RECIST version 1.0.
Time Frame: Tumour assessments were performed at baseline (tumour assessment obtained within 4 weeks prior to beginning of treatment), week 8, and every 8 weeks thereafter.
Population: Treated set (TS). TS consisted of all patients who were dispensed study medication and have taken at least 1 dose of Afatinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 41
Percentage of participants | 2 [0 to 13]

2. Secondary Outcome: Percentage of Participants With Disease Control (DC)
Description: Percentage of participants with OR or stable disease (SD) as determined by RECIST version 1.0.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 41
Percentage of participants | 59 [42 to 74]

3. Secondary Outcome: Progression Free Survival (PFS) Time
Description: PFS time defined as time from the start of treatment to the earliest of progression (RECIST), clinical progression (investigator), start of new anti-cancer treatment or death.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 41
Weeks | 15.86 [8.14 to 19.14]

4. Secondary Outcome: Summary of Pre-dose Concentrations of Afatnib in Plasma
Description: Pre-dose Concentrations of Afatinib in Plasma at Steady State on Days 15, 29 and 57 (Cpre,ss,15, Cpre,ss,29 and Cpre,ss,57)
Time Frame: Day 15, 29 and 57
Population: Patients with no data available for the relevant parameter and dose were excluded from analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 30
ng/mL
  Cpre,ss,15 (N=13) | 35.0 (74.9)
  Cpre,ss,29 (N=12) | 22.6 (79.5)
  Cpre,ss,57 (N=5) | 27.9 (96.1)

ADVERSE EVENTS:
Time Frame: First administration of trial medication until 28 days after last administration of trial medication
Arm/Group | Afatinib 50mg
Serious Adverse Events (participants affected / at risk) | 19/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 50mg (N=41)
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Pancreatitis acute (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 1
General physical health deterioration (General disorders) | 4
Pyrexia (General disorders) | 1
Spinal pain (General disorders) | 1
Bacterial infection (Infections and infestations) | 1
Clostridium colitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia klebsiella (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Spinal column injury (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Epilepsy (Nervous system disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 50mg (N=41)
Blepharitis (Eye disorders) | 5
Conjunctivitis (Eye disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 36
Dyspepsia (Gastrointestinal disorders) | 3
Mouth ulceration (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 11
Stomatitis (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 12
Asthenia (General disorders) | 12
Chest pain (General disorders) | 5
Fatigue (General disorders) | 10
Mucosal inflammation (General disorders) | 7
Oedema peripheral (General disorders) | 4
Pain (General disorders) | 3
Pyrexia (General disorders) | 7
Bronchitis (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 6
Paronychia (Infections and infestations) | 8
Urinary tract infection (Infections and infestations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 22
Hypokalaemia (Metabolism and nutrition disorders) | 4
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Acne (Skin and subcutaneous tissue disorders) | 10
Alopecia (Skin and subcutaneous tissue disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 5
Erythema (Skin and subcutaneous tissue disorders) | 4
Intertrigo (Skin and subcutaneous tissue disorders) | 3
Nail disorder (Skin and subcutaneous tissue disorders) | 5
Nail toxicity (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 28
Skin fissures (Skin and subcutaneous tissue disorders) | 5
Skin lesion (Skin and subcutaneous tissue disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.